CLINICAL TRIAL: NCT06907537
Title: A Study to Verify the Sleep-improving Effects of the Test Food Consumption: a Randomized, Placebo-controlled, Double-blind, Parallel-group Comparison Study
Brief Title: A Study to Verify the Sleep-improving Effects of the Test Food Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthomedico Inc. (Other)
Collaborators: AOBA KASEI CO., LTD. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 04400-0010-16; UMIN000057422 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2025-03-27; First posted 2025-04-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-05

CONDITIONS: Healthy Japanese
Keywords: Plasmalogen; Sleep condition
MeSH Terms: interventions — Food; Plasmalogens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasmalogen (Active Comparator): Take 1 mg/day of plasmalogen
  Interventions: Dietary Supplement: Food containing plasmalogen
- Placebo (Placebo Comparator): Take 0 mg/day of plasmalogen
  Interventions: Dietary Supplement: Food without plasmalogen

INTERVENTIONS:
Dietary Supplement: Food containing plasmalogen — Take four capsules per day in the morning.
  Arms: Plasmalogen
Dietary Supplement: Food without plasmalogen — Take four capsules per day in the morning.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test in Japanese adults who feel sleepy when they wake up. The question it aims to answer are:

•Does taking plasmalogens reduce sleepiness upon waking?

Participants will be given the following tasks:

* Take 4 capsules daily containing plasmalogens for 12 weeks.
* Answer the questionnaire on sleepiness1 when they wake up.
* Answer the questionnaire on daytime sleepiness2. Researchers will compare plasmalogens and placebo groups to see if plasmalogens reduce sleepiness upon waking.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese
2. Men or women
3. Adults
4. Healthy individuals
5. Individuals whose Zc score of "sleepiness on rising" is relatively low at screening

Exclusion Criteria:

1. Individuals who are undergoing medical treatment or have a medical history of malignant tumor, heart failure, or myocardial infarction
2. Individuals who have a pacemaker or an implantable cardioverter defibrillator (ICD)
3. Individuals who are currently undergoing treatment of any of the following chronic diseases: cardiac arrhythmia, liver disorder, chronic kidney disease, cerebrovascular disorder, rheumatic disease, diabetes mellitus, dyslipidemia, hypertension, or any other chronic diseases
4. Individuals who are undergoing medical treatment or have a medical history of any of the following diseases: mental disorders (e.g., depression), sleep apnea syndrome, hypersomnia, narcolepsy, insomnia, or valvular heart disease
5. Individuals who have habits of consuming foods or using devices to improve sleep
6. Individuals who have irregular sleeping habits due to lifestyle such as night shifts
7. Individuals who fall under the following sleeping conditions: sleeping in the same room with two or more people, living with preschool-aged children, living with individuals who require nursing care, or having their sleep potentially disturbed by the influence of others
8. Individuals who have nocturia two times or more
9. Individuals who usually drink to excess (average of more than about 20 g/day as absolute alcohol intake) {500 mL: a medium bottle of beer or about 1.5 cans of canned chu-hi, 180 mL: 1 go of sake or about 1.5 glasses of wine, 90 mL: half-go with shochu, 60 mL: a glass of whiskey brandy (double)}
10. Individuals who are taking "Foods for Specified Health Uses" or "Foods with Functional Claims"
11. Individuals who are taking medications (including herbal medicines) or supplements
12. Individuals who are allergic to medicines or foods related to the test product, or have a gelatin allergy or sea squirt-induced asthma
13. Individuals who are pregnant, lactating, or planning to become pregnant during this study
14. Individuals who have been enrolled in other clinical studies within the last 28 days before the agreement to participate in this study or plan to participate in another study during this study
15. Individuals who are judged as ineligible to participate in this study by the physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
The measured value of Zc score of "sleepiness on rising" in the OSA sleep inventory MA version (OSA-MA) after the 12-week intervention | After the 12-week intervention
  The OSA-MA is used to assess sleep quality. Individuals are asked to complete the questionnaire immediately after waking on the examination day and two days before the examination. The raw scores from each examination day will be converted to Zc scores, and the three-day mean, rounded to one decimal place, will be used as the measured value. "Sleepiness on rising" consists of four questions. Higher score indicates better outcome.

SECONDARY OUTCOMES:
The measured value of Zc score of "sleepiness on rising" in the OSA-MA after the 6-week intervention | After the 6-week intervention
  The OSA-MA is used to assess sleep quality. Individuals are asked to complete the questionnaire immediately after waking on the examination day and two days before the examination. The raw scores from each examination day will be converted to Zc scores, and the three-day mean, rounded to one decimal place, will be used as the measured value. "Sleepiness on rising" consists of four questions. Higher score indicates better outcome.
The measured values of Zc score of "initiation and maintenance of sleep," "frequent dreaming," "refreshing," and "sleep length" in the OSA-MA after the 6 and12-week intervention | After the 6 and12-week intervention
  The OSA-MA is used to assess sleep quality. Individuals are asked to complete the questionnaire immediately after waking on the examination day and two days before the examination. The raw scores from each examination day will be converted to Zc scores, and the three-day mean, rounded to one decimal place, will be used as the measured value. "Initiation and maintenance of sleep" consists of five questions, "frequent dreaming" consists of two questions, "refreshing" consists of three questions, and "sleep length" consists of two questions. Higher scores indicate better outcomes.
The measured value of total score of the Athens Insomnia Scale (AIS) after the 6 and12-week intervention | After the 6 and12-week intervention
  The AIS is used to assess sleep-related issues over the past month. Individuals are asked to answer eight sleep-related questions by selecting one of four response options, indicating experiences they have had at least three times per week in the past month. Lower score indicates better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tsuyoshi Takara, MD, Study Chair — Medical Corporation Seishinkai, Takara Clinic
Locations (2):
- Japan (2):
  - Nerima Medical Association Minami-machi Clinic, Nerima-ku, Tokyo
  - Medical Corporation Seishinkai, Takara Clinic, Shinagawa-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No
Data sharing will be discussed among the research affiliates after the study is completed.